CLINICAL TRIAL: NCT00875732
Title: CHOosing the rIght paCing Mode in Heart failurE : Should Heart Failure Patients With Bradycardia Receive Biventricular Pacemakers Rather Than Conventional Pacemakers?
Brief Title: Choosing the Right Pacing Mode in Heart Failure - The CHOICE Trial
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chest, Heart and Stroke Association Scotland (Other); Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, AChoy, Dr. Anna Maria Choy, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELD001
Record Dates: First submitted 2009-03-31; First posted 2009-04-03 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
Keywords: Resynchronization; Device; Bradycardia; atrioventricular block; Cardiac Resynchronization
MeSH Terms: conditions — Heart Failure; Bradycardia; Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Biventricular Pacing
  Interventions: Device: Bi Ventricular Pacing
- 2 (Active Comparator): Right Ventricular Pacing
  Interventions: Device: Right Ventricular Pacing

INTERVENTIONS:
Device: Bi Ventricular Pacing
  Arms: 1
Device: Right Ventricular Pacing
  Arms: 2

SUMMARY:
The aim of the study is to see if biventricular pacemakers offer any advantage over conventional pacemakers in patients with heart failure who require pacemakers. The endpoints will be the 6 minute walking distance along with markers of cardiovascular function.

The investigators' hypothesis is that biventricular pacing is preferable to conventional pacing in these heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

1. Left ventricular systolic dysfunction.
2. Atrio-ventricular node disease.
3. Anticipated to be more than 40% paced, (including patients in permanent atrial fibrillation).
4. Ability to walk independently (walking aid permitted).

Exclusion Criteria:

1. Patients meeting criteria for CRT by current guidelines will be excluded.
2. Life expectancy less than12 months.
3. Inability to walk independently.
4. Patients not likely to be compliant with follow-up.
5. Bradyarrhythmia due with sino-atrial disease only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
6 minute hall walk test | Baseline, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Endothelial Function | Baseline, 3, 6, 9 and 12 months
Cardiac Output | Baseline, 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ninewells Hospital & Medical School, Dundee, UK, United Kingdom